CLINICAL TRIAL: NCT03162458
Title: Multicenter Double-blind Placebo-controlled Parallel Group Randomized Clinical Trial of Efficacy and Safety of Anaferon for Children Liquid Dosage Form in the Treatment of Acute Upper Respiratory Infections
Brief Title: Clinical Trial of Efficacy and Safety of Anaferon for Children Liquid Dosage Form in the Treatment of Acute Upper Respiratory Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-AD-006
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Results first posted 2018-08-03 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Acute Upper Respiratory Infections
MeSH Terms: interventions — anaferon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaferon for children (Experimental)
  Interventions: Drug: Anaferon for children (liquid dosage form)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (liquid dosage form)

INTERVENTIONS:
Drug: Anaferon for children (liquid dosage form) — 10 drops per dose. Day 1: 10 drops every 30 minutes for the first 2 hours, followed by three more doses regularly spaced during the rest of the day. Day 2 to 5: 10 drops three times daily.
  Arms: Anaferon for children
Drug: Placebo (liquid dosage form) — 10 drops per dose. Day 1: 10 drops every 30 minutes for the first 2 hours, followed by three more doses regularly spaced during the rest of the day. Day 2 to 5: 10 drops three times daily.
  Arms: Placebo

SUMMARY:
Purpose of the study:

* To assess efficacy of Anaferon for children liquid dosage form in the treatment of acute upper respiratory tract infections.
* To assess safety of Anaferon for children liquid dosage form in the treatment of acute upper respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged 1 month to 3 years.
2. Diagnosis of acute upper respiratory infection based on a doctor's examination of the patient: body temperature at least 37.8°C when visiting a doctor + symptom scores ≥3 (presence of at least 1 general symptom and 1 nasal/ throat/chest symptom).
3. The first 24 hours from the beginning of manifestations of acute upper respiratory infection.
4. Acute respiratory viral infections season.
5. The possibility to start treatment within 24 hours of the onset of acute upper respiratory infection symptoms.
6. Availability of a patient information sheet (Informed Consent form) signed by the patient's parents/adopters to confirm the child's participation in the clinical trial signed by one parent/adopter of patient.

Exclusion Criteria:

1. Suspected pneumonia or bacterial infection or the presence of a disease requiring usage of antibacterial drugs starting from day 1 of the illness onset.
2. Clinical symptoms of severe influenza/ARI (acute respiratory infection) requiring hospitalization.
3. Suspected early manifestations of diseases that have symptoms similar to ARI symptoms (other infectious diseases, influenza-like syndrome at the onset of systemic connective tissue disorders, hematologic neoplasms and other pathology).
4. Documented (prior diagnosis) or suspected disease such as

   * primary or secondary immunodeficiency: а) lymphoid immunodeficiency (T-cell and/or B-cell immunity, immunodeficiencies with predominant antibody deficit, b) phagocyte deficits; c) complement factor deficit; d) combined immunodeficiency including AIDS secondary to HIV infection; toxic, autoimmune, infectious, or radial panleukopenia syndrome; general lymphocytopenia syndrome; syndrome of lymphocyte polyclonal activation; postsplenectomia syndrome; congenital asplenia; syndrome of immune complexes pathology associated with infectious, autoimmune and allergic diseases;
   * cystic fibrosis, primary ciliary dyskinesia, bronchopulmonary dysplasia, congenital malformations of the respiratory system, including malformations of upper respiratory tract, and other chronic lung disease;
   * malignant neoplasm.
5. Exacerbation or decompensation of chronic diseases affecting ability to participate in the clinical study.
6. Medical history of polyvalent allergy.
7. Allergy/ intolerance to any of the components of medications used in the treatment.
8. Use of medications listed in 'Prohibited concomitant treatments/medications' within 2 weeks before study entry.
9. Drug use or alcohol use (more than 2 alc. units daily) by the patient's parent(s)/adopter(s).
10. Mental disorders of patient's parent(s)/adopter(s).
11. Patients whose parents/adopters, from the investigator's point of view, will fail to comply with the observation requirements of the trial or with the intake regimen of the investigated medicines.
12. Participation in other clinical studies in the course of 3 months (or 1-2 months for infants under two months of age) prior to the inclusion in the trial.
13. Patient's parents/adopters are related to the clinical trial site's research staff directly involved in the trial or are the immediate family member of the researcher. The immediate family members include husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
14. The patient's parent/adopter works for OOO "NPF "MATERIA MEDICA HOLDING" (i.e., the company's employee, part-time employee under contract or appointed official in charge of the trial, or their immediate family).

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2015-04-29 (Actual); Study Completion 2015-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - LLC Center for Vaccine Prevention "DIAVAKS", Moscow
  - Municipal Health Care Institution "City Child Health Clinical Polyclinic №5", Perm
  - St. Petersburg State Budgetary Health Care Institution "Сity Polyclinic №44", Saint Petersburg
  - St. Petersburg State Health Care Institution "Children's City Polyclinic No. 45 Nevsky District", Saint Petersburg
  - Alliance Biomedical-Russian Group LLC, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "Children's City Hospital No. 22", Saint Petersburg
  - Federal State Budgetary Educational Institutionof Higher Education "Yaroslavl State Medical University" of the Ministry of Healthcare of the Russian Federation, Yaroslavl

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anaferon for Children | Placebo
Started | 71 | 71
Completed | 71 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaferon for Children | Placebo | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.8 (1.0) | 1.9 (1.0) | 1.9 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 35 | 39 | 74
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 71 | 71 | 142

OUTCOME MEASURES:

1. Primary Outcome: Average Illness Duration (the Interval Between the Start of the Trial Treatment and the Time When Recovery/Improvement - Based on Patient Diary Data)
Description: based on patient diary data
Time Frame: From the time of randomization until the time of recovery/improvement, assessed up to 14 days
Population: Intention to treat set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
hours | 87.7 (31.5) | 103.3 (19.4)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Severity of the Disease Within 5 Days Was Assessed Using the "Area Under the Curve" for the Total Symptom Score (TSS) at 1-5 Days (According to the Diary of the Patient).
Description: The TSS was based on the severity of each of acute upper respiratory tract infection (URTI) symptom.
  The TSS includes 11 symptoms: Body temperature / fever, Non-specific URTI symptoms (Decreased activity / Malaise, Impaired appetite / refusal of feeding, Painful appearance, Sleep disturbance) and Nose /Throat symptoms (Runny nose, Nasal congestion, Sneezing, Hoarseness, Sore throat, Cough).
  The severity of each URTI symptom was scored on a symptom severity scale (0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms).
  Minimum score=0; maximum score=33. The severity of URTI symptoms was recorded by one of the patient's parents/adopter on a diary card twice a day (morning and evening) on Days 1-5.
Time Frame: On days 1-5 of observation
Population: Intention to treat set
Measure: Mean (Standard Deviation); unit: AUC score*day
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
AUC score*day | 25.6 (17.2) | 33.6 (17.7)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.0004, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Patients With Recovery on Days 2, 3, 4 and 5 of Observation (Based on Patient Diary Data)
Description: based on patient diary data
Time Frame: On Days 2-5 of the treatment
Population: Intention to treat set
Measure: Number; unit: percentage of participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
percentage of participants
  Day 2 | 9.9 | 0
  Day 3 | 29.6 | 4.2
  Day 4 | 39.4 | 18.3
  Day 5 | 64.8 | 57.8
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.055, Log Rank

4. Secondary Outcome: Average Duration of Fever (i.e. Body Temperature >37.3°С)
Description: based on patient diary data
Time Frame: From the time of randomization until the time of normal body temperature, assessed up to 14 days
Population: Intention to treat set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
hours | 47.3 (30.3) | 57.0 (31.6)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.051, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Mean Body Temperatures, Measured in the Morning and Evening on Days 2-5 (Based on Patient Diary Data)
Description: based on patient diary data
Time Frame: On Days 2-5 of the treatment
Population: Intention to treat set
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
°C
  Day 2, Morning | 37.4 (0.7) | 37.6 (0.7)
  Day 3, Morning | 37.0 (0.6) | 37.1 (0.5)
  Day 4, Morning | 36.9 (0.6) | 36.9 (0.4)
  Day 5, Morning | 36.7 (0.5) | 36.7 (0.6)
  Day 2, Evening | 37.4 (0.8) | 37.5 (0.8)
  Day 3, Evening | 37.1 (0.7) | 37.1 (0.6)
  Day 4, Evening | 36.9 (0.6) | 36.9 (0.6)
  Day 5, Evening | 36.7 (0.3) | 36.8 (0.5)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Mean body temperatures, measured in the morning on Days 2-5 (based on patient diary data); Test type: Superiority; p = 0.19, ANOVA
Statistical Analysis 2: Comparison: Anaferon for Children vs Placebo; Mean body temperatures, measured in the evening on Days 2-5 (based on patient diary data); Test type: Superiority; p = 0.44, ANOVA

6. Secondary Outcome: Percentage of Patients With Body Temperature ≤37.30С on Days 2-5 of Observation
Description: based on patient diary data
Time Frame: On Days 2-5 of observation
Population: Intention to treat set
Measure: Number; unit: percentage of participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
percentage of participants
  Day 2 | 28.2 | 12.7
  Day 3 | 56.3 | 43.7
  Day 4 | 73.2 | 74.7
  Day 5 | 88.7 | 83.1
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.15, Log Rank

7. Secondary Outcome: Total Symptom Score on Days 3 and 6 of Observation Based on the Results of Pediatrician's Examination
Description: The Total Symptom Score (TSS) was based on the severity of each of acute upper respiratory tract infection (URTI) symptom.
  The TSS includes 11 symptoms: Body temperature / fever, Non-specific URTI symptoms (Decreased activity / Malaise, Impaired appetite / refusal of feeding, Painful appearance, Sleep disturbance) and Nose /Throat symptoms (Runny nose, Nasal congestion, Sneezing, Hoarseness, Sore throat, Cough).
  The severity of each URTI symptom was scored on a symptom severity scale (0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms).
  Minimum score=0; maximum score=33. The severity of URTI symptoms was recorded by the study researchers (pediatricians) on the case record form on Days 1, 3, 6.
Time Frame: On Days 1, 3, 6 of the treatment
Population: Intention to treat set
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
Score
  Day 1 | 11.8 (3.9) | 12.5 (4.6)
  Day 3 | 6.0 (4.7) | 8.0 (4.6)
  Day 6 | 1.9 (2.7) | 2.8 (4.8)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.004, ANOVA

8. Secondary Outcome: Severity of the Disease Within 5 Days Was Assessed Using the "Area Under the Curve" for the Total Symptom Score (TSS) on Days 1, 3, 6 (According to the Results of Pediatrician's Examination)
Description: The TSS was based on the severity of each of acute upper respiratory tract infection (URTI) symptom.
  The TSS includes 11 symptoms: Body temperature / fever, Non-specific URTI symptoms (Decreased activity / Malaise, Impaired appetite / refusal of feeding, Painful appearance, Sleep disturbance) and Nose /Throat symptoms (Runny nose, Nasal congestion, Sneezing, Hoarseness, Sore throat, Cough).
  The severity of each URTI symptom was scored on a symptom severity scale (0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms).
  Minimum score=0; maximum score=33. The severity of URTI symptoms was recorded by the study researchers (pediatricians) on the case record form on Days 1, 3, 6.
Time Frame: on Days 1, 3, 6
Population: Intention to treat set
Measure: Mean (Standard Deviation); unit: AUC score*day
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
AUC score*day | 12.6 (7.0) | 16.0 (7.6)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Number of Antipyretic Use (for Prescribed Indications) on Days 1-5 of Treatment (Based on Patient Diary Data)
Description: based on patient diary data
Time Frame: on Days 1-5 of treatment
Population: Intention to treat set
Measure: Mean (Standard Deviation); unit: Number of intakes
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
Number of intakes
  Day 1 | 0.8 (0.9) | 0.7 (0.9)
  Day 2 | 0.5 (1.1) | 0.5 (0.8)
  Day 3 | 0.2 (0.7) | 0.2 (0.5)
  Day 4 | 0.2 (0.7) | 0.1 (0.5)
  Day 5 | 0.1 (0.3) | 0.1 (0.4)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.63, ANOVA

10. Secondary Outcome: Percentage of Patients With Complications of Illness, Including Those Requiring Antibiotic Administration or Hospitalization) for 14 Days of Observation
Time Frame: From the time of randomization up to 14 days
Population: Intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 71 | 71
percentage of participants | 2.8 | 4.2
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered from Day 1 to Day 14
Description: Adverse/Serious adverse events were registered in patients of the Full Analysis Set (n=142, Safety Population)
Arm/Group | Anaferon for Children | Placebo
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 7/71 | 4/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaferon for Children (N=71) | Placebo (N=71)
Hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Herpes Labialis (Infections and infestations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Administration related reaction (Immune system disorders) | 1 (1) | 0 (0)
Eustachitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Rhinitis purulent (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Daytime sleepiness (Nervous system disorders) | 0 (0) | 1 (1)
Purulent conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Right otitis media (acute, non-suppurative) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Bilateral otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other